CLINICAL TRIAL: NCT06087679
Title: The SongDanceT1 Study: Stress, Ongoing Self- Monitoring and Diabetes, Nerve Stimulation and Cognitive Empowerment. An Implementation Study Combined With an Observer-blinded Randomized Controlled Interventional Trial (SongDance T1D)
Brief Title: The SongDanceT1 Study: Stress, Ongoing Self- Monitoring and Diabetes, Nerve Stimulation and Cognitive Empowerment.
Acronym: SongDanceT1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Steno Diabetes Center Copenhagen (Other)
Collaborators: Department of Medicine, Endocrine Unit Herlev University Hospital, Herlev, Denmark (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 72976
Record Dates: First submitted 2021-07-07; First posted 2023-10-18 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Autonomic Dysfunction; Stress, Psychological
MeSH Terms: conditions — Primary Dysautonomias; Stress, Psychological

STUDY DESIGN:
Intervention Model Description: Single-center parallel placebo-controlled randomized trial
Who Masked: Care Provider
Masking Description: The participants are randomized 1/1: active/control, and a person, who has no direct contact to the participants, performs the randomization. The study is open to the participating participants and the instructors of the active group. The study is blinded to all others, including the statisticians who make the main analyses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Selfcare program (Experimental): 6-month intervention period with a PPS guided selfcare based intervention program
  Interventions: Behavioral: PPS guided selfcare based intervention program
- Control group (No Intervention): Treatment as usual

INTERVENTIONS:
Behavioral: PPS guided selfcare based intervention program — Guided selfcare programme (Please refer to project description)
  Other Names: ULLCARE
  Arms: Selfcare program

SUMMARY:
In an implementation study, designed as a RCT in people with type 1 diabetes(T1D) and an elevated Pressure pain sensitivity of the chest bone(PPS) as indicative of dysfunction of the autonomic nervous system (ANSD), to describe the effect of a selfcare programe on the following outcome measures:

1. PPS, and the effect on health risk factors associated to quality of life, physiology and metabolism.

   People acceptance of the program: Can T1D people comply with the program and integrate the program into their daily life?
2. The professional staff acceptance of the program: Does the staff comply to the program and does the program comply to the routines of the clinical department?

DETAILED DESCRIPTION:
Type 1 Diabetes is a chronic disease, affecting mostly young people and associated with depression among approx. 20-25% of the people.

Depression in T1D is further associated with a poor treatment adherence, hyperglycemia, increased health costs, increased complications, cognitive decline, and also increased all-cause and coronary heart disease mortality.

Besides the 3 classical complications to T1D, retinopathy, nephropathy and neuropathy, dysfunction of the autonomic nervous system (ANSD) is often seen, and is regarded as a complication to long standing T1D. The latter is typically tested as impairment of autonomic control of the cardiovascular system and is designated cardiac autonomic neuropathy (CAN). The prevalence is approx. 15% of definite ANSD (higher when including incipient ANSD) and depending on the duration of the diabetes disease.

Autonomic nervous system dysfunction is in general associated to chronic stress, depression, and reduced quality of life (QOL). In people with ischemic heart disease (IHD), it is associated to increased morbidity and mortality. In T1D, ANSD is associated with increased morbidity, especially cardiovascular disease, kidney disease and peripheral neuropathy.

Pressure pain sensitivity of the chest bone (PPS), usually measured by a special algometer (StressMeter), was originally found to be associated to acute and chronic stress. However, recent studies have found a close association between chronic stress and ANSD, linking these two together (for review see www.stressmeter.org). PPS seems to measure primarily sympathetic autonomic function, probably in the brain, and potentially at the level of the lateral hypothalamus. As such, resting PPS seems to be indicative of autonomic function.

The PPS measurement device can be used by both professionals and people, and a non-pharmacological intervention, the ULLCARE®program, has been developed, with the ability to restore and maintain normal PPS. Simultaneously to a normalization in PPS, measures of autonomic function also seem to normalize. The key elements of this program are: 1) daily cognitive reflection based on the PPS measure as a behavioural guide for stress; 2) cutaneous sensory nerve stimulation with the aim to reduce an elevated PPS or maintain a low PPS, and 3) ongoing internet based professional surveillance with the aim to pro-actively intervene in the case of deviating or missing PPS measurements.

The concept to measure PPS and take action by aiming at reducing an elevated PPS and thus reduce the ANSD in chronic disease is thus established. The scientific background for the PPS measurement, the effects from reducing an elevated PPS, as well as the association to ANSD is presented on a research webpage: www.stressmeter.org

Research questions of the RCT study:

1. Does a simple individualized self-care -ased intervention program, that uses daily PPS measure as a feedback marker of the state of ANSD and fluctuations of stress, and followed by cutaneous sensory nerve stimulation reduce the elevated PPS?
2. If so, is this reduction associated with: (i) autonomic dysfunction restoration (as measured by: (i): improved CAN score test for the group of participants who have an elevated CAN score test at baseline; (ii) increase in the PPS response to tilting (ii) reduction of depression score, clinical stress score, neuropathic pain, and increase of QOL and empowerment?
3. Do T1D participants who respond to the intervention by a reduction of reduction of PPS ≥ 15 arbitrary units (i.e. responders; from the active and control group, alike) have a significant clinical effect, in terms of the included outcome measures, when comparing responders with non-responders?
4. Do people with type 1 diabetes have been exposed to situations/conditions in their lives, just around the time of the onset of their diabetes, which may indicate massive stress/ANSD?
5. If the PPS-measure is compared to Perceived stress scale (PSS), do we see a relevant association connection and similarly when comparing the Clinical stress sign score (CSS) and PSS?

Sub studies:

The study includes two separate sub studies. 3. Design A prospective, randomized observer-blinded controlled trial in which the effect of a 6-month intervention period with a PPS guided selfcare based intervention program (ULLCARE) + treatment as usual (TAU) (i.e. active group) is compared to a control group, who receives TAU.

In order to obtain an even distribution between the active group and the control group with respect to CAN score and glycated hemoglobin (HbA1c), the participants are stratified during the randomization procedure (see point 3.1) The study takes place at Steno Diabetes Centre Copenhagen (SDCC) but with the possibility that some or all parts of the active groups program can take place either virtually or in a private medical clinic.

With respect to this aim, a separate registration of the study will be submitted to The Danish Medicines Agency for approval. The documents for submission as well as for approval will be forwarded separately to the Scientific Ethics Committee.

The participants are randomized 1/1: active/control, and a person, who has no direct contact to the participants, performs the randomization. The study is open to the participating participants and the instructors of the active group. The study is blinded to all others, including the statisticians who make the main analyses. The personnel conducting the clinical examinations does not have access to the documents containing information about the treatment or treatment procedures. This is to prevent bias in the comparison between the treatment groups.

The participants are stratified in three groups depending on the CAN score obtained from the reflex tests obtained by the Vagus test: 1) CAN score = 0 (no autonomic neuropathy); 2) CAN score = 1 (borderline autonomic neuropathy); 3) CAN score ≥2 (definite autonomic neuropathy), and similarly in two groups with respect to HbA1c = 60 mmol/mol as discrimination value.

120 participants recruited from The Diabetic Neuropathy Screening Study (The DANES study) will be included in the trial, 60 in the active group and 60 in the control group. The DANES study is an ongoing study performed at SDCC, which is approved by the local ethical committee.

Inclusion criteria

* Diagnosed T1D
* BMI < 40
* PPS ≥ 60 arbitrary units (normal range: 30 - 60)
* Age < 75 years; age ≥ 18 years
* Manage the Danish language for proper use of instructions,
* Actively accepting to conduct a minimum of 20 minutes of self-care daily according to the ULLCARE program.

Exclusion criteria

* Use of Beta blockade medication, and tricyclic anti-depressive medication
* Previously diagnosed and treated for a psychiatric disorder, except for depression.
* A chronic competing disorder that statistically is life-shortening (such as advanced cancer with metastases).
* A chronic competing disorder that is not heart disease and not a diabetes co-morbidity, which clearly impairs the participant's QOL /e.g. COPD, cancer, chronic pain syndrome).
* People who cannot conduct the selfcare program (example: having one arm, only?

Flow of the inclusion process The initial contact to the study group is related to the DANES study, in which the participants are recruited from.

The first contact will be the one of the following two: (i) when the participant is examined as part of the DANES Study baseline examination, he or she will receive an invitation letter with respect to participate in the present study. If the participant wants to, next step is a meeting with a Songdance T1D researcher; (ii) for the participant for whom the initial DANES examination has been conducted and who at that examination had an elevated PPS, an invitation letter is send - similar to the one, which is used for the first mentioned group For the first Songdance meeting, the participant is recommended to bring an assessor. Prior to this meeting the following documents are send to the participant, allowing a minimum of 24 hours for reading the documents: 1) "Deltagerinformation, 2) "Samtykke erklæring", 3) "Forsøgspersoners rettigheder i et sundhedsvidenskabeligt forskningsprojekt" (version marts 2019), og 4) "før du beslutter dig". For this consultation, there will be emphasis on the fact that the information session is about a query of participation. The subject's right not to receive information on his/her health condition and disposition to disease will be reviewed and respected.

Secondly, if the participant wants to participate, the "Samtykke erklæring" must be returned to the study staff, preferable within a week after the information consult. Thereafter, the participant is scheduled for baseline examination.

Outcome measures Change after 6 months

1. Primary effect variable:

   Resting PPS
2. Secondary effect variables:

   Physiological measures:

   Total CAN score (Vagus) The three individual CAN score tests (reflex tests) Resting heart rate variability indices (HRV) Resting pulse, blood pressure PPS and cardiovascular response to a tilt table test Questionnaire derived outcome measures of quality of life
3. Tertiary effect variables:

Number of sick leave days (for people at work) Total number of elevated health risk factors; se below HbA1c Total insulin dose Insulin sensitivity estimated by daily insulin use (IE) divided by body weight. Urine Albumin/creatinine ratio BMI Serum lipids Kidney function measured as creatinine

Practical course

* The recruitment and thus the initial screening is among participants in the Danes Study (see section 4.4for details).
* The participation is 6 months for each participant (i.e. for the active group this is 6 months are first session)
* The inclusion period for the study is expected to be 6 months.
* All participants undergo examination at start, and after 6 months
* The following data are obtained:

  * Demografic data at baseline
  * Physiological data: resting PPS, Vagus, pulse rate and blood pressure
  * Questionnaires of life quality
* At the baseline visit patients are randomised to active or control follow up, by an independent person
* Participants in the active group receive the ULLCARE educational program®, are educated in PPS measurement for home use, and are followed by a professional coach, who conducts ongoing internet PPS measurement surveillance on a weekly basis.
* Persons in the control group (TAU) follow regular visits in the clinic as planned and are examined again at visit 2.

Methods 8.1 PPS measurement A StressMeter® (UllCare A/S, Hellerup, Denmark) is used, which is a scientifically validated, non-invasive and CE marked instrument (see www.stressmeter.org), developed to measure the /activity of the sympathetic autonomic nervous system by measuring the pressure pain sensitivity of the most painful point on the sternum between costa 3 to 5. The point is identified by finger pressure. After 10 minutes of rest in the supine position, the participant first learns his/hers pain threshold as the instructor applies a gradually increasing pressure over 5 sec. with the instrument, and the participant is instructed to say stop when the threshold of pain/discomfort is reached. If the instructor observes a noxious withdrawal reflex (i.e. an involuntary muscle contraction of the muscles around the eyes, the neck or upper limb) before the participant says stop, the procedure is stopped, and the PPS value is recorded. The instrument displays a number on a scale from 30 (corresponding to a pressure of 5 kg/cm2) to 100 (corresponding to a pressure of 0.5 kg/cm2), where an increased sensibility is accompanied by an increasing measure, meaning that a high PPS measure reflects a high level of stress (high sensitivity or low pain threshold). ANSD is defined as an elevated resting PPS measure ≥ 60 arbitrary units). A responder of an intervention, with the aim to reduce an elevated resting PPS, and thus ANSD, is defined as a reduction of resting PPS ≥ 15 arbitrary units; a non-responder is defined as a person who do not obtain such reduction.

The StressMeter has the following special features:

* Hidden measurement value until the measurement is completed.
* A calculation of the sensitivity to a tenderness score on a logarithmic scale similar to the decibel scale used to estimate the limit values of sound pressure in connection with a hearing test.
* An alarm that is activated by a pressure before the occurrence of any injury.
* A special foot pad that prevents irritation of the skin and which ensures that it is the pressure sensitivity of the periosteum that is measured and not that of the skin.

The UllCare program (assigned ULLCARE):

The basic elements of the intervention provided to the active group are as follows:

1. A self-care part.
2. A professional instruction in the PPS measurement, cognitive reflection in relation to the measure and nerve stimulation.
3. Continuous recording of the participants' PPS measurements through a web journal.

PPS measurement

The participants are instructed to perform the PPS measurement twice daily, similarly and as a supplement to the home blood glucose measurement. It is explained that:

* The PPS measure represents a simple measure for ANS function and the level of stress, but also for a variety of important diabetes and cardiovascular health risk factors, including HbA1c, blood pressure, heart rate, work of the heart, serum lipids, low grade inflammation, QOL, depression and persistent stress.
* All of these risk factors may improve concomitantly (if elevated) when PPS is persistently reduced to a level below 60 arbitrary units and with the ultimate goal to obtain a morning PPS below 45 arbitrary units.
* The present PPS guided self-care based non-pharmacological intervention will do the job when applied on a daily basis, similarly to daily tooth brushing for caries prevention.

Cutaneous sensory nerve stimulation:

The participants are instructed to perform the preventive nerve stimulation twice a day, plus ad hoc when they urgently want to reduce their stress. Nerve stimulation is done by applying pressure with a finger for one minute - one should feel it, but it should not cause any pain. This is done at the following acupuncture points: On the sternum at the level of the fourth intercostal space, and on the back, 3.8 cm lateral to the spinal process of the fourth and fifth thoracic vertebra. Nerve stimulation is done successfully, when the participant can observe that the tenderness of the point has been reduced after applying pressure for 20 to max 60 seconds. If this result has not been achieved, the patient is instructed to repeat the treatment on another tender point.

8.3 Blood and urine analyses Routine blood samples (HbA1c, creatinine and lipids) and a spot-urine sample (for the measurement of urinary albumin/creatinine ratio) are taken as part of the study at baseline and after 6 months. HbA1c is taken as part of routine work-up of the participant.

If the participant gives signed informed consent, a spare blood sample for future research purposes will be obtained at baseline and at 6 months visit and stored in a biobank.

Questionnaires

The following questionnaires will be included as outcome measures:

1. Diabetes empowerment is measured by the questionnaire DES-SF (Andersen RM et al, 2003)
2. Major depression inventory (MDI) (Bech P, 2012)
3. WHO-5 quality of life score (Bech P, 2012)
4. Clinical stress sign score (CSS) (Ballegaard S 2012, Bergmann N 2013; Axelsson A, 2014)
5. Perceived stress scale (PSS) (D'Alonzo KT 2019)
6. Epworth Sleepiness score (Chasen ER et al. 2013) + special designed questionnaire with focus on sleep disturbance
7. Diabetes treatment satisfaction questionnaire (Baccoro F et al, 2016)
8. Implementation study questionnaire according the WHO guide lines (Peter DH, 2013)
9. Problem Areas In Diabetes (PAID-20) (Polonsky WH et al. 1995)

Other measures

1. BMI: will be measured as weight in kilogram divided with height in meters squared.
2. Blood Pressure (mm Hg) and pulse (beats/minute): measured automatically conducted in the supine position after 10 minutes of rest (Thuasne automatic oscillometric blood pressure monitor) with an appropriate cuff size.
3. Work of the heart is measured as Pressure-Rate-Product (mm Hg/beats per minute: systolic blood pressure x heart rate).
4. ANS measures (conducted in the following order and initiated by 10 minutes of rest in the supine position:

   * PPS as described above
   * Tilt table test: the participant is passively tilted to 70 degrees upright position. PPS, pulse rate and blood pressure are recorded at: (i) end of the 10 minutes of rest, (ii) right after tilting (approximately one minute, and (iii) after being in the upright passive position for 7 minutes.
   * CAN score measured by Vagus® instrument (non-invasive procedure). This is a validated and CE labelled product (Vagus ®, Medicus Engineering Aps, Århus, Denmark). By non-invasive means, and after 10 minutes of rest, it includes resting heart rate plus a CAN score: beat-to-beat variation during three ANS stimulation tests conducted in the following order: 1) stand-up (tilting) (measures primarily sympathetic nervous activity), 2) deep breathing (measures primarily parasympathetic nervous activity), and 3) Valsalva maneuver (measures a combination of sympathetic and parasympathetic nervous activity). ANSD is defined by age-adjusted nomograms provided by the manufacturer. CAN score 0: no positive CAN score tests, which indicates no cardiac autonomic neuropathy (CAN); CAN score 1: one of the three tests is positive, which indicates borderline CAN; CAN score 2: two or more of the three tests are positive, which indicates definitive CAN.

Statistics Calculation of sample size and power analysis Calculation of sample size is based on the followed premises with respect to PPS: The Minimal Important Difference is 15 arbitrary units, mean PPS at baseline is estimated to be 75 arbitrary units, and with standard deviation 18. In a previous study of heart patients this result was achieved in 61% of the active group and 27% of the control group (OR 4,1, p<0,001) (Ballegaard et al. 2015). In a similar study in diabetes type 2 patients corresponding success rate was 67% and 28% respectively (OR 5,2, p<0,001). Based on these results we estimated the succesrate in the present study as 60% and 25% respectively. Alfa: 5, Beta: 80 %. Based on this we will include 60 participants in each group. We will include 120 participants in total. (https://biostat.app.vumc.org/wiki/Main/PowerSampleSize, version 3, 2014).

Cohens effect size (Cohen J 1994 is a fraction that consists of the difference in PPS from before intervention till after treatment for the active group, minus the same difference for the control group divided by the spread (i.e. standard deviation) of the change in PPS, when taking all participants together. Example: the PPS in the active group changes from 75 to 55 (75-55) = 20 a.u., while the PPS for the control group changes from 75 to 70 (75-70) = 5 a.u. This change in PPS is 20-5 = 15; if the spread on the PPS for all participants is 18, the effect size will be 15/18 = 0.8 Minimal clinically relevant effect size: 0.3 (Bech 1912).

Analysis of the effect variables Analyses of effect variables will be performed after 6 months. The associations between determinants and outcome measures will be estimated by using complete-case regression models adjusting for relevant confounders including age, sex and diabetes duration. Logistic regression analyses will be used for binary outcomes. Linear regression analyses will be used for continuous outcomes. Outcome variables will be log-transformed using the natural logarithm to meet model assumptions of the distribution of the model residuals if necessary. Interactions between sex and all determinants will be investigated in all models to investigate possible sex interactions differences. A level of significance of 5% will be used.

Analyses will be performed using SAS version 9.3(SAS Institute, Cary, NC).

Monitoring will be conducted by an independent Clinical Research Organization (CRO). If accepted the GCP unit of RegionHovedstaden (placed at Bispebjerg Hospital) will perform this monitoring.

The assigned CRO shall conduct study site monitoring to ensure that the human subject protection, study procedures and data collection processes are of high quality and meet the requirements and regulatory guidelines.

The designee will visit the site to install the equipment and perform a site initiation visit. To ensure that the study is conducted in accordance with the approved protocol, in compliance with GCP and applicable regulatory requirements, monitoring visits will be performed by the appointed CRO monitor in accordance to the monitoring plan.

When the study is complete, the study monitorshall make a close-out visit to the study site.

The patient samples are planned to be collected during ordered blood draws and thus no adverse events are anticipated. Any unanticipated adverse device effects noted with the use of the analyzer in the laboratory or the point of care site shall be reported immediately to the sponsor of the study, who will inform Ull Care.

Both positive, inconclusive and negative results will be compiled in one or more scientific articles and sent to international peer-reviewed publications regarding publication. Collaborators will be co-authors in accordance to the Vancouver recommendation for authorship.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed T1D
* BMI < 40
* PPS ≥ 60 arbitrary units (normal range: 30 - 60)
* Age < 75 years; age ≥ 18 years
* Manage the Danish language for proper use of instructions,
* Actively accepting to conduct a minimum of 20 minutes of self-care daily according to the ULLCARE program.

Exclusion Criteria:

* Use of Beta blockade medication, and tricyclic anti-depressive medication
* Previously diagnosed and treated for a psychiatric disorder, except for depression.
* A chronic competing disorder that statistically is life-shortening (such as advanced cancer with metastases).
* A chronic competing disorder that is not heart disease and not a diabetes co-morbidity, which clearly impairs the participant's QOL /e.g. COPD, cancer, chronic pain syndrome).
* People who cannot conduct the selfcare program (example: having one arm, only)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-07-08 (Actual); Primary Completion 2024-01-30 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
change in resting PPS | Measured at baseline and 6-months follow-up
  A StressMeter® (UllCare A/S, Hellerup, Denmark) is a device that measure the ammount of pressure applied to the skin. Participants will apply presure on specific pressure point (describe in the project description) and read an abitrary number of pressure og a display when dyscomfort is felt.

SECONDARY OUTCOMES:
Total CAN score (Vagus®) | Measured at baseline and 6-months follow-up
  CAN score measured by Vagus® instrument (non-invasive procedure). This is a validated and CE labelled product (Vagus ®, Medicus Engineering Aps, Århus, Denmark). By non-invasive means, and after 10 minutes of rest, it includes resting heart rate plus a CAN score: beat-to-beat variation during three ANS stimulation tests (CARTS) conducted in the following order: 1) stand-up (tilting) (measures primarily sympathetic nervous activity), 2) deep breathing (measures primarily parasympathetic nervous activity), and 3) Valsalva maneuver (measures a combination of sympathetic and parasympathetic nervous activity). ANSD is defined by age-adjusted nomograms provided by the manufacturer (Fleischer et al 2015). CAN score 0: no positive CAN score tests, which indicates no cardiac autonomic neuropathy (CAN); CAN score 1: one of the three tests is positive, which indicates borderline CAN; CAN score 2: two or more of the three tests are positive, which indicates definitive CAN.
The three individual CAN score tests (CARTs) | Measured at baseline and 6-months follow-up
  CAN score measured by Vagus® instrument (non-invasive procedure). This is a validated and CE labelled product (Vagus ®, Medicus Engineering Aps, Århus, Denmark). By non-invasive means, and after 10 minutes of rest, it includes resting heart rate plus a CAN score: beat-to-beat variation during three ANS stimulation tests (CARTS) conducted in the following order: 1) stand-up (tilting) (measures primarily sympathetic nervous activity), 2) deep breathing (measures primarily parasympathetic nervous activity), and 3) Valsalva maneuver (measures a combination of sympathetic and parasympathetic nervous activity). ANSD is defined by age-adjusted nomograms provided by the manufacturer (Fleischer et al 2015). CAN score 0: no positive CAN score tests, which indicates no cardiac autonomic neuropathy (CAN); CAN score 1: one of the three tests is positive, which indicates borderline CAN; CAN score 2: two or more of the three tests are positive, which indicates definitive CAN.
Resting heart rate variability indices (HRV) | Measured at baseline and 6-months follow-up
  HRV measures willl be analyzed from 5-minute resting heart rate recording from the Vagus device
Resting pulse | Measured at baseline and 6-months follow-up
  Resting measures willl be analyzed from 5-minute resting heart rate recording from the Vagus device
Resting Blood pressure | Measured at baseline and 6-months follow-up
  mesured after five minutes of rest and calculated as the mean of two consecutive measures with the cuff on a healthy arm with the patient in a sitting position using automated oscillometric device.
  blood pressure recorders were used
cardiovascular response to a tilt table test | Measured at baseline and 6-months follow-up
  • Tilt table test: the participant is passively tilted to 70 degrees upright position. pulse rate and blood pressure are recorded at: (i) end of the 10 minutes of rest, (ii) right after tilting (approximately one minute, and (iii) after being in the upright passive position for 7 minutes
PPS response to a tilt table test | Measured at baseline and 6-months follow-up
  * PPS as described above
  * Tilt table test: the participant is passively tilted to 70 degrees upright position. PPS are recorded at: (i) end of the 10 minutes of rest, (ii) right after tilting (approximately one minute, and (iii) after being in the upright passive position for 7 minutes.
diabetes empowerment, measured by the questionnaire DES-SF | Measured at baseline and 6-months follow-up
  Mannually filled out by participants. Evaluated as a total score of the questionnaire
Major depression inventory (MDI) | Measured at baseline and 6-months follow-up
  Mannually filled out by participants. Evaluated as a total score of the questionnaire
WHO-5 quality of life score | Measured at baseline and 6-months follow-up
  Mannually filled out by participants. Evaluated as a total score of the questionnaire
Clinical stress sign score (CSS) | Measured at baseline and 6-months follow-up
  Mannually filled out by participants. Evaluated as a total score of the questionnaire
Epworth Sleepiness score | Measured at baseline and 6-months follow-up
  Mannually filled out by participants. Evaluated as a total score of the sleep quality from the questionnaire
special designed questionnaire with focus on sleep disturbance | Measured at baseline and 6-months follow-up
  Mannually filled out by participants. Evaluated as a total score of the sleep quality from the questionnaire
Diabetes treatment satisfaction questionnaire (DTSQ) | Measured at baseline and 6-months follow-up
  Mannually filled out by participants. Evaluated as a total score of the questionnaire
Implementation study questionnaire according the WHO guidelines | Measured at baseline and 6-months follow-up
  Mannually filled out by participants. Evaluated as a total score of the questionnaire
Problem Areas In Diabetes (PAID-20) | Measured at baseline and 6-months follow-up
  Mannually filled out by participants. Evaluated as a total score of the questionnaire

OTHER OUTCOMES:
Number of sick leave days (for people at work) | Number of sick days between baseline and 6-months follow-up
  Repported by participants
Total number of elevated health risk factors | Measured at baseline and 6-months follow-up
  Discrimination values for each outcome measure will be as follows:
  HbA1c: ≥ 53 mmol/mol Total cholesterol: ≥ 5.0 mmol/L LDL cholesterol: ≥ 3.5 mmol/L HDL cholesterol: ≤ 0.9 mmol/L Triglyceride: ≥ 2.0 mmol/L CAN score: ≥ 1 PPS: ≥ 60 arbitrary units Blood pressure: ≥ 130/85 mm Hg (i.e. systolic BP ≥ 135 or diastolic BP ≥ 85 mmHg (supine BP after 10 minutes of rest in the supine position) Heart rate: ≥ 70 beats/minute PRP: ≥ 10.000 mmHg/beats per minute BMI: ≥ 25 kg/m2 Depression score: MDI ≥ 15 WHO 5: score < 50 Clinical stress score: ≥ 8
  A reduction of the total number of elevated risk factors (maximum number: 14) will be used as a success criterium.
HbA1c | Measured at baseline and 6-months follow-up
  serum samples analyzed by high performance liquid chromatography.
Total insulin dose | Logged at baseline and 6-months follow-up
  Repported by participants
Insulin sensitivity | Logged and measured at baseline and 6-months follow-up
  Estimated by daily insulin use (IE) divided by body weight.
Urine Albumin/creatinine ratio | Measured at baseline and 6-months follow-up
  Spot urine samples af Urine Albumin/creatinine ratio analyzed by quantitative immunological turbidimetry
BMI | Measured at baseline and 6-months follow-up
  Measured by height and weight
Serum lipids | Measured at baseline and 6-months follow-up
  Total cholesterole, LDL, HDL and triglycerides analyzed by standard enzymatic colorimetry techniques
Kidney function measured as creatinine | Measured at baseline and 6-months follow-up
  Serum creatinine analyzed by quantitative immunological turbidimetry

CONTACTS AND LOCATIONS:
Locations (1):
- Steno Diabetes Center Copenhagen, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: No
Anonymized data will be made available on reasonable request.